CLINICAL TRIAL: NCT00864539
Title: The Prevalence of Vitamin D Insufficiency in Primary School Children and Comparison of the Effect of Calcium-Vitamin D-Fortified Milk, -Orange Juice and Calcium-Vitamin D Supplement
Brief Title: Comparison of the Efficacy of Calcium-cholecalciferol Foodstuffs and Calcium-cholecalciferol Supplement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Tirang R. Neyestani, associate professor, National Nutrition and Food Technology Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P/25/47/2027
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Vitamin D Status; Healthy
Keywords: vitamin D fortification; milk; orange juice; supplement; efficacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- fortified milk (Experimental): daily intake of milk fortified with 100 IU vitamin D and 500 mg calcium/200 mL
  Interventions: Dietary Supplement: fortified milk
- plain milk (Active Comparator): daily intake of 200 mL plain milk
  Interventions: Dietary Supplement: plain milk
- fortified orange juice (Experimental): daily intake of orange juice fortified with 100 IU vitamin D and 500 mg calcium
  Interventions: Dietary Supplement: fortified orange juice
- plane juice (Active Comparator): subjects receiving plain orange juice
  Interventions: Dietary Supplement: plain orange juice
- vitamin D-Ca supplement (Experimental): Subjects receiving daily supplement containing 500 mg + 200 IU vitamin D
  Interventions: Dietary Supplement: calcium-vitamin D supplement
- Placebo (Placebo Comparator): Subjects receiving daily placebo containing 1g starch
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fortified milk — daily intake of milk fortified with 100 IU vitamin D and 500 mg calcium/200 ml package for 10 weeks
  Other Names: FM
  Arms: fortified milk
Dietary Supplement: plain milk — daily intake of 200 ml plain milk
  Other Names: PM
  Arms: plain milk
Dietary Supplement: fortified orange juice — daily intake of orange juice fortified with 100 IU vitamin D and 500 mg calcium/250 ml package
  Other Names: FJ
  Arms: fortified orange juice
Dietary Supplement: plain orange juice — daily intake of 250 ml plain orange juice
  Other Names: PJ
  Arms: plane juice
Dietary Supplement: calcium-vitamin D supplement — daily calcium-vitamin D supplement (500 mg calcium + 200 IU vitamin D)
  Other Names: SP
  Arms: vitamin D-Ca supplement
Dietary Supplement: Placebo — daily placebo
  Other Names: PL
  Arms: Placebo

SUMMARY:
This study is conducted in two phases. At the first phase, the prevalence of vitamin D insufficiency in primary school-children in Tehran is determined during the cold seasons of 2008. Then, the efficacy of calcium-vitamin D-fortified milk, -orange juice and supplement is compared in six selected primary schools.

DETAILED DESCRIPTION:
At the first step, serum 25-(OH)D, PTH(parathyroid hormone), osteocalcin, bone alkaline phosphatase, calcium, phosphorous, and magnesium is evaluated. Anthropometric and dietary intake data is also collected. In the second phase, we have 6 experimental groups: (1) plain milk; (2) calcium-vitamin D-fortified milk (containing 500 mg Ca and 100 IU vitamin D/200 mL package); (3) plain orange juice; (4) fortified orange juice containing equal amounts of calcium and vitamin D as fortified milk; (5) calcium-vitamin D supplement (500 mg calcium and 200 IU vitamin D); and (6) placebo. Each group consists of 40-60 children (9-11 years) from both sexes. All above-mentioned biochemical, anthropometric and dietary intake data is collected both in the beginning and in the end of interventional period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 9-11 years
* Being healthy (no apparent clinical disease)
* Informed consent signed by child's parent(s)

Exclusion Criteria:

* Subjects receiving vitamin D, calcium or omega-3 supplement
* Unwillingness to continue the study
* Subjects with type 1 diabetes, allergy, kidney disorders

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 585 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, Ph.D., Study Chair — National Nutrition and Food Technology Research Institute, P.O. Box 19295-4741

RESULTS

PARTICIPANT FLOW:
Groups:
- Fortified Milk: daily intake of milk fortified with 100 IU vitamin D and 500 mg calcium/200mL
- Plain Juice: subjects receiving plain orange juice
- Vitamin D-Calcium Supplement: Subjects receiving daily supplement containing 500 mg + 200 IU vitamin D
- Placebo: Subjects receiving daily placebo containing 1 g starch
Period: Overall Study
Arm/Group | Fortified Milk | Plain Milk | Fortified Orange Juice | Plain Juice | Vitamin D-Calcium Supplement | Placebo
Started | 104 | 95 | 102 | 96 | 103 | 85
Completed | 95 (Attrition was due to absence or unwillingness to donate blood.) | 72 (Attrition was due to absence or unwillingness to donate blood.) | 92 (Attrition was due to absence or unwillingness to donate blood.) | 89 (Attrition was due to absence or unwillingness to donate blood.) | 81 (Attrition was due to absence or unwillingness to donate blood.) | 71 (Attrition was due to absence or unwillingness to donate blood.)
Not Completed | 9 | 23 | 10 | 7 | 22 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fortified Milk | Plain Milk | Fortified Orange Juice | Plain Juice | Vitamin D-Calcium Supplement | Placebo | Total
Number analyzed (Participants) | 104 | 95 | 102 | 96 | 103 | 85 | 585
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 104 | 95 | 102 | 96 | 103 | 85 | 585
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.3 (0.7) | 10.1 (0.8) | 10.1 (0.6) | 9.9 (0.8) | 10.4 (0.6) | 9.8 (0.8) | 10.1 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 50 | 48 | 65 | 79 | 59 | 352
  Male | 53 | 45 | 54 | 31 | 24 | 26 | 233
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 104 | 95 | 102 | 96 | 103 | 85 | 585
Serum levels of 25(OH)D [Mean (Standard Deviation); unit: nmol/L] — Anthropometric and laboratory assessments were carried out at the beginning and at the end of the intervention. In order to perform blood analyses, 3mL of venous blood was taken from all the participants. Laboratory tests included hemoglobin, hematocrit, serum levels of 25(OH)D, iPTH, osteocalcin, bone-specific alkaline phosphatase (BAP), calcium, phosphorous, magnesium, total protein and albumin.
  nmol/L | 30.5 (24.7) | 25.0 (17.2) | 18.0 (14.4) | 26.6 (22.0) | 16.6 (17.8) | 19.6 (23.7) | 23.0 (20.9)

OUTCOME MEASURES:

1. Primary Outcome: Serum Levels of 25hydroxy Vitamin D(25(OH)D)Compared to the Due Control Group
Description: Serum level of 25(OH)D was determined using competitive protein binding assay (CPBA) method.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Fortified Milk | Plain Milk | Fortified Orange Juice | Plain Juice | Vitamin D-Calcium Supplement | Placebo
Number analyzed (Participants) | 104 | 95 | 102 | 96 | 103 | 85
nmol/L | 21.6 (16.6) | 21.2 (17.0) | 33.3 (27.6) | 31.5 (34.0) | 26.0 (24.3) | 21.8 (28.2)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Fortified Milk | Plain Milk | Fortified Orange Juice | Plain Juice | Vitamin D-Calcium Supplement | Placebo
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/95 | 0/102 | 0/96 | 0/103 | 0/85
Other Adverse Events (participants affected / at risk) | 0/104 | 0/95 | 0/102 | 0/96 | 0/103 | 0/85

LIMITATIONS AND CAVEATS:
Because of very cold winter, it was not possible to extend the intervention period to 12 weeks or longer. Moreover, it was impossible to fortify the foodstuffs with more than 50% of RDA(recommended daily allowance) because of legal problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes